CLINICAL TRIAL: NCT04157244
Title: The Feasibility of a Tailored Music Intervention to Reduce Symptoms of Sleep Disruption in Older Adults With Dementia
Brief Title: The Music, Sleep and Dementia Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Darina Petrovsky, PhD, RN, Postdoctoral Research Fellow, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 829256
Record Dates: First submitted 2019-10-07; First posted 2019-11-08 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Dementia; Alzheimer Disease; Circadian Rhythm Disorders; Circadian Rhythm Sleep Disorder; Insomnia; Hypersomnia; Cognitive Impairment; Cognitive Decline; Mild Cognitive Impairment; Frontotemporal Dementia; Neurocognitive Disorders; Vascular Dementia; Sleep Disorder; Memory Impairment
MeSH Terms: conditions — Dementia; Alzheimer Disease; Chronobiology Disorders; Sleep Disorders, Circadian Rhythm; Sleep Initiation and Maintenance Disorders; Disorders of Excessive Somnolence; Cognitive Dysfunction; Frontotemporal Dementia; Neurocognitive Disorders; Dementia, Vascular; Sleep Wake Disorders; Memory Disorders

STUDY DESIGN:
Intervention Model Description: Wait-list controlled design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Tailored Music (Experimental): 4-week tailored music listening intervention delivered to persons with dementia and their caregivers via a tablet.
  Interventions: Behavioral: Tailored music listening intervention
- 4-week Wait-list control (No Intervention): 4-week wait-list control (Note: participants will be crossed over to 4-week tailored music listening intervention delivered to persons with dementia and their caregivers via a tablet)

INTERVENTIONS:
Behavioral: Tailored music listening intervention — The music intervention consists of listening to preferred soothing music at bedtime for 30 minutes every night for four weeks (28 sessions total). This theory based caregiver-assisted intervention builds on the evidence-based protocol of using individualized music to decrease agitation in nursing home residents. It also accounts for sleep-inducing properties of music.
  Arms: Experimental: Tailored Music

SUMMARY:
The specific aims of this studyare to examine the 1) feasibility; 2) acceptability; and 3) preliminary efficacy of a tailored music intervention in home-dwelling older adults with dementia suffering from sleep disruption. Sixty dyads (older adults with dementia and their caregivers) will be randomized to receive the tailored music intervention immediately or following a four week delay.

DETAILED DESCRIPTION:
Sleep disruption in older adults living with Alzheimer's disease and related dementias (ADRD) is very debilitating and contributes to increased institutionalization, reduced cognitive function, and accelerated disease progression. Furthermore, sleep disruption is linked to poor health outcomes in caregivers (CGs), such as poor quality of life and increased CG burden. Given the potential harmful side effects of pharmacologic treatment, non-pharmacologic approaches, such as music, may provide a safer alternative to reducing sleep disruption in this vulnerable population. Listening to music has been shown to decrease agitation, anxiety and depression in nursing home residents with ADRD. A growing body of literature suggests that individualized music may improve sleep quality in older adults with early memory loss, but its efficacy has not been demonstrated in older adults with ADRD in the community, where most older adults with ADRD live. If proven feasible and acceptable, tailored music interventions can then be tested for efficacy in reducing sleep disruption.

Music selections will be individualized to older adults with ADRD and account for known sleep-inducing properties. Feasibility of processes that are key to the success of the subsequent study will be examined. Preliminary efficacy of the intervention will be assessed using objective (actigraphy) and subjective (proxy reported) sleep quality measures. In addition, qualitative data will be solicited from the dyads examining the acceptability and satisfaction with the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 and older
* Physician diagnosis of probable ADRD using standard assessments and diagnostic criteria
* Presence of sleep problems determined first during phone screening using NPI sleep disorders item, then using proxy-rated Sleep Disorders Inventory (SDI) (presence of at least one sleep disturbance symptom of moderate severity)
* Stable dose of psychotropic medications, sedatives/hypnotics, anti-dementia or opioids in the past 90 days (typical time frame in clinical trials) prior to enrollment to minimize confounding effects of medications
* Tolerates and agrees to wear wrist actigraph
* Responsive to their environment (e.g., able to understand short commands)
* Sufficient English to complete questionnaires

Exclusion Criteria:

* Planned transition to another residential or institutional care setting in less than 3 months
* Hearing impairment (defined as inability to hear a normal speaking voice at a distance of 1-1/2 feet)
* Presence of extrapyramidal symptoms affecting non-dominant hand which may include persons with the following diagnoses: schizophrenia, bipolar disorder, Huntington's disease, Parkinson's disease, Lewy Body dementia due to REM sleep disorders
* Currently enrolled in an interventional clinical trial for ADRD aimed to improve sleep
* Acute sleep disruption within 2 weeks of screening as it may indicate sleep disorders not related to ADRD or delirium
* End stage disease (i.e. cancer, bed bound)

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-03-12 (Actual); Primary Completion 2021-01-12 (Actual); Study Completion 2021-01-12 (Actual)

PRIMARY OUTCOMES:
Study Measures Completion | Baseline
  Number of participants who complete study measures in accordance with protocol schedule of events
Study Measures Completion | 4 weeks
  Number of participants who complete study measures in accordance with protocol schedule of events
Acceptability of the study components | 4 weeks
  Two questions from a survey developed by Gitlin and colleagues (2010) which examines satisfaction with participation and perceived benefits.
  The survey uses a scale of 1-3 (1- Not at all to 3-A great deal) to rate caregiver perceived 1) overall benefit from participating in the study and 2) improvement in life of person's with dementia.
  Min score 2, maximum score 6 (with higher scores indicating greater satisfaction and perceived benefits)

SECONDARY OUTCOMES:
Objective sleep measures | 4 weeks
  Measured using an actigraphy bracelet worn by person with dementia for consecutive 24-hour periods for 4 weeks. The actigraph will measure: 1) Sleep latency (Time it takes a person to fall asleep starting from first intention to sleep); 2) Wake after sleep onset (Time awake during the night, beginning from the time person falls asleep); 3) Total sleep duration (Actual time person is asleep)
The Quality of Life in Alzheimer's Disease Scale (QOL-AD) | Baseline and 4 weeks
  Person with dementia quality of life. The QOL-AD scale uses a scale of 1-4 (poor, fair, good, or excellent) to rate a variety of life domains, including the patient's physical health, mood, relationships, activities, and ability to complete tasks.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gitlin LN, Winter L, Dennis MP, Hodgson N, Hauck WW. Targeting and managing behavioral symptoms in individuals with dementia: a randomized trial of a nonpharmacological intervention. J Am Geriatr Soc. 2010 Aug;58(8):1465-74. doi: 10.1111/j.1532-5415.2010.02971.x. Epub 2010 Jul 19. PMID 20662955
- [Background] Gitlin LN, Winter L, Dennis MP, Hodgson N, Hauck WW. A biobehavioral home-based intervention and the well-being of patients with dementia and their caregivers: the COPE randomized trial. JAMA. 2010 Sep 1;304(9):983-91. doi: 10.1001/jama.2010.1253. PMID 20810376
- [Derived] Petrovsky DV, Bradt J, McPhillips MV, Sefcik JS, Gitlin LN, Hodgson NA. Tailored Music Listening in Persons With Dementia: A Feasibility Randomized Clinical Trial. Am J Alzheimers Dis Other Demen. 2023 Jan-Dec;38:15333175231186728. doi: 10.1177/15333175231186728. PMID 37470678
- [Derived] Jespersen KV, Pando-Naude V, Koenig J, Jennum P, Vuust P. Listening to music for insomnia in adults. Cochrane Database Syst Rev. 2022 Aug 24;8(8):CD010459. doi: 10.1002/14651858.CD010459.pub3. PMID 36000763